CLINICAL TRIAL: NCT02019160
Title: Effectiveness of Biannual Application of Silver Nitrate Solution Followed by Sodium Fluoride Varnish in Arresting Early Childhood Caries in Preschool Children: a 30-month, Randomised, Double-blind, Non-inferiority Trial
Brief Title: Effectiveness of Dental Caries Arrest Treatment in Primary Teeth Using AgNO3 Followed by NaF Varnish
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chun-Hung Chu, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: chuch14
Record Dates: First submitted 2013-12-11; First posted 2013-12-24 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Early Childhood Caries
Keywords: silver nitrate; sodium fluoride; silver diamine fluoride; caries; non-inferiority trial
MeSH Terms: interventions — Silver Nitrate; Sodium Fluoride; silver diamine fluoride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Silver nitrate (Experimental): Biannual application of 25% AgNO3 solution followed by 5% NaF varnish.
  Interventions: Drug: 25% AgNO3 solution followed by 5% NaF varnish
- Silver diamine fluoride (Active Comparator): Biannual application of 38% SDF solution followed by placebo varnish.
  Interventions: Drug: 38% SDF solution followed by placebo varnish

INTERVENTIONS:
Drug: 25% AgNO3 solution followed by 5% NaF varnish — Dosage of 4.4μg±1.4μg fluoride per use
  Other Names: silver nitrate; sodium fluoride
  Arms: Silver nitrate
Drug: 38% SDF solution followed by placebo varnish — Dosage of 8.8μg±2.8μg fluoride per use
  Other Names: silver diamine fluoride
  Arms: Silver diamine fluoride

SUMMARY:
* Aim: This randomised controlled trial will systematically compare the efficacy of a 25% AgNO3 solution followed by 5% NaF varnish with that of a 38% SDF solution in arresting caries teeth among preschool children when applied at half-yearly intervals over a 30-month period.
* Method: The extension of the Consolidated Standards of Reporting Trials 2010 Statement will be followed for this 30-month, randomised, double-blinded, non-inferiority clinical trial. Approximately 2,400 kindergarten children will be screened and at least 826 children with caries will be recruited. This sample size is sufficient for an appropriate statistical analysis (power at 90% [β=0.10] with a 2-sided type-I error of α=0.05), allowing for a 18% drop-out rate. The children will be randomly allocated into 2 groups to treat their caries over a 30-month period: Group A - biannual application of a 25% AgNO3 solution followed by a 5% NaF varnish, and Group B - biannual application of a 38% SDF solution followed by a placebo varnish.Clinical examinations will be conducted at 6-month intervals to assess whether the caries are arrested. Information on confounding factors such as oral hygiene habits will be collected through a parental questionnaire.
* Possible results and implications: As the first of its kind, this study would help to determine whether AgNO3 followed by NaF is at least as effective as SDF in arresting childhood caries. If so, because 25% AgNO3 and 5% NaF contain less silver and fluoride, respectively, than 38% SDF, their use would be more favourable than SDF in young children.

ELIGIBILITY:
Inclusion Criteria:

* Kindergarteners who have joined our outreach dental service will be invited to join this study. Preschool children aged 3-4 years who have tooth decay and are attending the first year of kindergarten will be invited to join this study.

Exclusion Criteria:

* Children who are uncooperative and difficult to manage, have major systemic diseases, or are on long-term medication will be excluded.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1070 (Actual)
Dates: Start 2014-09; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
The hardness of cavity on tooth by probing | The follow-up oral examinations will be conducted every 6 months for 30 months totally
  We expect that topical application of 25% AgNO3 solution followed by 5% NaF varnish and of 38% SDF solution can both effectively arrest ECC.

CONTACTS AND LOCATIONS:
Overall Officials: Chun Hung Chu, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, China

REFERENCES:
- [Background] Braga MM, Mendes FM, De Benedetto MS, Imparato JC. Effect of silver diammine fluoride on incipient caries lesions in erupting permanent first molars: a pilot study. J Dent Child (Chic). 2009 Jan-Apr;76(1):28-33. PMID 19341576
- [Background] Chu CH, Fung DS, Lo EC. Dental caries status of preschool children in Hong Kong. Br Dent J. 1999 Dec 11;187(11):616-20; discussion 605. doi: 10.1038/sj.bdj.4800347. PMID 16163284
- [Background] Chu CH. Treatment of early childhood caries: a review and case report. Gen Dent. 2000 Mar-Apr;48(2):142-8. PMID 11199573
- [Background] Chu CH, Lo EC, Lin HC. Effectiveness of silver diamine fluoride and sodium fluoride varnish in arresting dentin caries in Chinese pre-school children. J Dent Res. 2002 Nov;81(11):767-70. doi: 10.1177/0810767. PMID 12407092
- [Background] Chu CH, Lo EC. A review of sodium fluoride varnish. Gen Dent. 2006 Jul-Aug;54(4):247-53. PMID 16903196
- [Derived] Gao SS, Duangthip D, Wong MCM, Lo ECM, Chu CH. Randomized Trial of Silver Nitrate with Sodium Fluoride for Caries Arrest. JDR Clin Trans Res. 2019 Apr;4(2):126-134. doi: 10.1177/2380084418818482. Epub 2019 Feb 15. PMID 30931709
- [Derived] Chu CH, Gao SS, Li SK, Wong MC, Lo EC. The effectiveness of the biannual application of silver nitrate solution followed by sodium fluoride varnish in arresting early childhood caries in preschool children: study protocol for a randomised controlled trial. Trials. 2015 Sep 25;16:426. doi: 10.1186/s13063-015-0960-2. PMID 26407698